CLINICAL TRIAL: NCT07069972
Title: Comparing Efficacy and Safety of Telitacicept and Belimumab in Systemic Lupus Erythematosus: A Prospective Multicenter Cohort Study.
Brief Title: A Prospective Comparative Study Involving Multiple Units to Evaluate the Efficacy and Safety of Telitacicept and Belimumab in the Treatment of Systemic Lupus Erythematosus.
Status: Not yet recruiting | Type: Observational
Sponsor: Yipeng Liu (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); Affiliated Hospital of Shandong University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Yipeng Liu, Clinical Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2025(106)
Record Dates: First submitted 2025-06-13; First posted 2025-07-17 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Telitacicept; Belimumab; Efficacy and Safety
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- The Telitacicept group（the overall SLE population）: The participants in this group were diagnosed with SLE and were selected to use Telitacicept as the treatment drug.This study is an observational study and no active intervention is carried out.
- The Belimumab group（the overall SLE population）: The participants in this group were diagnosed with SLE and were selected to receive belimumab as the treatment drug.This study is an observational study and no active intervention is carried out.
- The Telitacicept group（the lupus nephritis subgroup）: The participants in this group were diagnosed with LN and were selected to receive telitacicept as the treatment drug.This study is an observational study and no active intervention is carried out.
- The Belimumab group（the lupus nephritis subgroup）: The participants in this group were diagnosed with LN and were selected to receive belimumab as the treatment drug.This study is an observational study and no active intervention is carried out.

SUMMARY:
The objective of this observational study is to compare the efficacy and safety of telitacicept versus belimumab in systemic lupus erythematosus (SLE) patients aged 18-65 years. The primary questions it aims to answer are:

* In the overall SLE population: What are the SRI-4 response rates for both drugs?
* In the lupus nephritis subgroup: What are the major renal response rates for both drugs?

Participants will autonomously select their treatment regimen (add-on telitacicept or belimumab) based on:

* The patient's objective clinical condition at enrollment
* Physician's assessment
* Joint decision-making between physicians and patients/family members As an observational study, no active intervention will be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18 - 65 years old;
* Meets the revised SLE classification criteria of the American College of Rheumatology in 1997 or the SLE diagnostic classification criteria issued by EULAR/ACR in 2019;
* The SELENA-SLEDAI score is at least 8 points (clinical symptoms are no less than 6 points, excluding positive anti-double-stranded DNA (anti-dsDNA) and low complement);
* Has not responded well to hormone and/or immunosuppressant treatment, is intolerant or has recurrence, and is willing to accept tixocortinib/belimumab as a therapeutic drug.

Exclusion Criteria:

* Any of the following conditions exists: active central nervous system disease, severe active lupus nephritis, HIV infection, hepatitis B or C virus infection, low gamma globulinemia, liver dysfunction;
* eGFR < 30 mL/min/1.73m², or undergoing hemodialysis or kidney transplantation;
* Pregnant women, or women who are about to become pregnant in the near future, or lactating women;
* Participants who are simultaneously participating in other clinical studies;
* Within 1 year before randomization, received B-cell targeted therapy (including belimumab);
* During treatment, used traditional Chinese medicine with immunosuppressive effects (such as Tripterygium wilfordii, White Peony Root, etc.) in combination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with systemic lupus erythematosus through clinical examination at the First Affiliated Hospital of Shandong First Medical University, the Affiliated Hospital of Shandong University of Traditional Chinese Medicine, and the People's Hospital of Wuhan University
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with a Systemic Lupus Erythematosus Response Index-4 (SRI-4) response(the overall SLE population) | From baseline to the end of 2-year treatment period
  1. A reduction of ≥ 4 points in the SELENA-SLEDAI score from baseline;
  2. And no new BILAG A-level organ or ≤ 2 new BILAG B-level organs compared to baseline;
  3. And no worsening in the physician's global assessment (PGA) (an increase of < 0.30 points from baseline).
The response rate for major kidney treatments(the lupus nephritis subgroup) | From baseline to the end of 2-year treatment period
  1. 24-hour urine PCR ≤ 0.7 g/g (70 mg/mmol);
  2. eGFR decline does not exceed 20% of the baseline or is ≥ 60 ml/min/1.73 m2;
  3. No rescue treatment was adopted due to treatment failure.

SECONDARY OUTCOMES:
Complete renal response rate(the lupus nephritis subgroup) | From baseline to the end of 2-year treatment period
  1. 24-hour urine PCR < 0.5 g/g (50 mg/mmol);
  2. Stable or improved renal function (not exceeding 10% - 15% of the baseline).
Proportion of Participants with Stable SLEDAI and PGA Scores(the overall SLE population) | From baseline to the end of 2-year treatment period
  The percentage of study participants whose SLEDAI score decreased by at least 4 points and whose PGA did not worsen.
The proportion of participants in the study who had their hormone dosage reduced(the overall SLE population) | From baseline to the end of 2-year treatment period
  The ratio of study participants whose prednisone dose was reduced by ≥25% or ≤7.5 mg/day compared to the baseline at 44-48 weeks.
The time of recurrence occurrence(the overall SLE population) | From baseline to the end of 2-year treatment period.
  The time of the first recurrence or the first severe recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No